CLINICAL TRIAL: NCT03673124
Title: A Phase II Trial of Ribociclib (LEE011) Plus Letrozole in Women With Recurrent Low-Grade Serous Carcinoma of the Ovary, Fallopian Tube or Peritoneum
Brief Title: Ribociclib and Letrozole Treatment in Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-3026
Record Dates: First submitted 2018-09-11; First posted 2018-09-17 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Low Grade Serous Carcinoma
Keywords: ovary; peritoneum; fallopian tube
MeSH Terms: conditions — Cystadenocarcinoma, Serous | interventions — ribociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ribociclib and letrozole (Other): Ribociclib 600mg oral daily for 3 weeks then 1 week off plus Letrozole 2.5 mg oral daily
  Interventions: Drug: Ribociclib; Drug: Letrozole

INTERVENTIONS:
Drug: Ribociclib — 600 mg by mouth daily for 21 days followed by 7 days off treatment
Drug: Letrozole — 2.5 mg by mouth daily

SUMMARY:
The study evaluates the response to treatment with Ribociclib and Letrozole in patients with low grade serous cancer of the ovary, fallopian tube or peritoneum.

DETAILED DESCRIPTION:
Ribociclib (formerly LEE011) is an orally bioavailable, highly selective small molecule inhibitor of cyclin-dependent kinases 4 and 6 (CDK4/6). Ribociclib has been approved by the United States Food and Drug Administration (U.S. FDA) and the European Commission as an initial endocrine-based therapy for the treatment of postmenopausal women with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative advanced or metastatic breast cancer in combination with an aromatase inhibitor based on a randomized, double-blind, placebo-controlled, international clinical trial (MONALEESA-2). Additional marketing authorizations are under review by health authorities. Additional phase III clinical trials for the treatment of hormone receptor positive (HR+) breast cancer patients, as well as several other phase I or II clinical studies are being conducted.

Letrozole is a highly potent, orally active non-steroidal competitive inhibitor of the aromatase enzyme system. It effectively inhibits the conversion of androgens to estrogens both in vitro and in vivo. It is indicated both as first-line treatment of postmenopausal women with hormone receptor positive or hormone receptor unknown locally advanced or metastatic breast cancer as well as for the treatment of advanced breast cancer in postmenopausal women with disease progression following antiestrogen therapy.

Based on encouraging results in women with advanced hormone-receptor-positive breast cancer, a clinical trial for women with recurrent low-grade serous carcinoma is warranted. Furthermore, such a trial would have great appeal to women with recurrent low-grade serous carcinoma, a cohort with limited therapeutic options. Although low-grade serous carcinoma is a rather uncommon histologic subtype, prolonged overall survival results in a relatively high prevalence.

ELIGIBILITY:
Patients eligible for inclusion in this study must meet all of the following criteria:

1. Patient has signed the Informed Consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements.
2. Age > 18 years at time of study entry.
3. Willingness and ability to comply with study and follow-up procedures.
4. Histological confirmation of diagnosis of low-grade serous carcinoma of ovary, fallopian tube or peritoneum; Original diagnosis of de novo low-grade serous carcinoma or Original diagnosis of serous borderline tumor with subsequent diagnosis of low-grade serous carcinoma.

   • In order to prevent inclusion of patients with high-grade serous carcinoma, diagnosis of low-grade serous carcinoma will be verified as part of screening review by a gynecologic pathologist. Tissue for confirmation can be from primary tumor or recurrence.
5. Patient must have recurrent, measurable disease by RECIST v1.1.
6. There are no restrictions on number of prior therapies.
7. Patient cannot have previously received a prior cyclin dependent kinase inhibitor (CDKi). Patients who were treated with letrozole or another aromatase inhibitor for other indications must have not taken the drug for 6 months prior to initiating letrozole for this trial and may not have progressed on treatment.
8. Patients must not have remaining ovarian function to be included. In women who have at least one retained ovary, menopause must be confirmed with laboratory confirmation. Women who have ovarian function are eligible but must be placed on hormonal suppression. Menopause must be confirmed with laboratory confirmation, to include an estradiol level as this is assessed within 8 weeks of patient having been on tamoxifen.
9. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
10. Resolution of all acute toxic effects of prior therapy or surgical procedures to National Cancer Institute (NCI) CTCAE Grade ≤ 1. Patients with grade 1 taxane-induced neuropathy, any grade alopecia, amenorrhea, or other toxicities not considered a safety risk for the patient as per investigator's discretion are eligible. 1. Patient has adequate bone marrow and organ function as defined by the following laboratory values at screening:

    * Absolute neutrophil count ≥1.5 × 109/L
    * Platelets ≥100 × 109/L
    * Hemoglobin ≥9.0 g/dL
    * Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
    * International Normalized Ration (INR) ≤1.5 (unless patient is receiving permitted anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug). Serum creatinine <1.5 mg/dL or creatinine clearance ≥50 mL/min
    * In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x Upper Limit of Normal (ULN). If the patient has liver metastases, ALT and AST <5 x ULN
    * Total bilirubin < ULN; or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome.

12. Patient with available standard 12-lead ECG with the following parameters at screening:

* QTcF interval at screening <450msec (using Fridericia's correction)
* Resting heart rate 50-90bpm 13. Must be able to swallow ribociclib and letrozole capsules/tablets. 14. Patients receiving tamoxifen or toremifene must have washout period of 5 half-lives prior to randomization.

Patients eligible for this study must not meet any of the following criteria:

1. Patient has a known hypersensitivity to any of the excipients of ribociclib or letrozole.
2. Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer. Patients with known brain metastases are excluded.
3. Patients with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

   * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
   * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases.
4. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
5. Patient has a known history of HIV infection (testing not mandatory).
6. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
7. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

   * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
   * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
   * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade Atrioventricular (AV) block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
   * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

     * Risk factors for Torsades de Pointe (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
     * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
     * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
     * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening
8. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug (see Table 1 for details):

   * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
   * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
   * Herbal preparations/medications, dietary supplements.
9. Participation in other studies involving investigational drug(s) within 30 days prior to randomization or within 5 half-lives of the investigational product (whichever is longer) or participation in any other type of medical research judged not to be scientifically or medically compatible with this study. If the patient is enrolled or planned to be enrolled in another study that does not involve an investigational drug, the agreement of Novartis study medical lead is required to establish eligibility.
10. Patient is currently receiving warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed. Direct-Acting Oral Anticoagulants (DOACS) are permitted.
11. Patient is currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment. The following uses of corticosteroids are permitted: a short duration (,5 days) of systemic corticosteroids; any durations of topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
12. Patient who has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥25% of the bone marrow (Ellis, 1961) was irradiated.
13. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
14. Patient with a Child-Pugh score B or C.
15. Patients who are pregnant or breastfeeding.
16. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 3 weeks after study drug discontinuation. Highly effective contraception methods include:

    * Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
17. Current use of food or drugs known to be potent CYP3A4 inhibitors, drugs known to be potent CYP3A4 inducers, and drugs that are known to prolong the QT interval unless the prohibited concomitant medication can be replaced by other drugs of less potential to inhibit or induce CYP3A4 or prolong QT interval (See Appendix C for Prohibited Concomitant Medications).
18. Patients whose tumors contain both low-grade serous carcinoma (LGSC) and high-grade serous carcinoma (HGSC)
19. Patients with history of haemopoietic stem cell or bone marrow transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Slomovitz, MD, Study Chair — GOG
Locations (27):
- United States (27):
  - University of California, San Francisco, San Francisco, California
  - UF Heath, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Saint Vincent Hospital and Health Care Center, Inc., Indianapolis, Indiana
  - St. Joseph Mercy Hospital Cancer Care Center, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Valley Hospital Inc., Ridgewood, New Jersey
  - New Mexico Cancer Care Alliance/University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates, Albuquerque, New Mexico
  - Miami Valley Hospital, Centerville, Ohio
  - The Ohio State Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Care Specialists and Research Institute , LLC, Tulsa, Oklahoma
  - Western Pennsylvania Hospital/West Penn Hospital, Pittsburgh, Pennsylvania
  - Abington Memorial Hospital, Willow Grove, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Parkland Health and Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center - Texas Medical Center, Houston, Texas
  - Houston Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 74 participants were screened for eligibility in the study. Out of these, 51 participants were determined to be eligible for enrollment. The recruitment period spanned from June 2018 to February of 2023.The first patient was enrolled on May 20, 2019.
Groups:
- Ribociclib and Letrozole: Ribociclib 600 mg administered orally daily for 21 days followed by 7 days off in 28-day treatment cycle in combination with Letrozole 2.5 mg administered orally daily for 28 days. Treatment continues until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ribociclib and Letrozole
Started (Enrolled and eligible) | 51
Completed (Eligible and treated) | 49
Not Completed | 2
Not completed — Eligible with no protocol therapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ribociclib and Letrozole
Number analyzed (Participants) | 49
Age, Customized [Count of Participants; unit: Participants]
  Age (Years): 20-29 | 4
  Age (Years): 30-39 | 6
  Age (Years): 40-49 | 7
  Age (Years): 50-59 | 8
  Age (Years): 60-69 | 17
  Age (Years): 70-79 | 6
  Age (Years): 80-89 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 3
  Race: White | 44
  Race: Unknown | 1
  Race: Declined to Report | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 9
  Ethnicity: Not Hispanic or Latino | 38
  Ethnicity: Declined to Report | 1
  Ethnicity: Unknown | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49
Performance Status (ECOG) [Count of Participants; unit: Participants] — ECOG 0 is fully active, able to carry on all pre-disease performance without restriction.
  ECOG 1 is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    ECOG 0 | 27
    ECOG 1 | 21
    Not Reported | 1
Site of Disease [Count of Participants; unit: Participants]
  Ovary | 44
  Peritoneum | 5
FIGO Stage at Diagnosis (ohr) [Count of Participants; unit: Participants] — FIGO stage at diagnosis was reported by each participant institution according to their standard practice. In general, a higher FIGO stage indicates more advanced disease.
  Participants
    I | 2
    II | 1
    III | 36
    IV | 9
    Not Reported | 1
Prior Surgery [Count of Participants; unit: Participants]
  No | 3
  Yes | 46
Prior Radiation Therapy (ohr) [Count of Participants; unit: Participants]
  No | 48
  Yes | 1
Any Prior Immunologic/Chemo/Hormonal/Biologic/Antiangiogenic/Other therapy [Count of Participants; unit: Participants]
  No | 3
  Yes | 46
Lines of Prior Therapy (ohr) [Count of Participants; unit: Participants] — Any immunologic/chemo/hormonal/biologic/antiangiogenic/other therapy reported by participation sites, where a line of therapy was defined by the participation sites' standards.
  Participants
    0 | 3
    1 | 20
    2 | 7
    3 | 6
    4 | 7
    5 | 1
    6 or more | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants in the analysis population who achieved a complete response or partial response, as assessed by RECIST 1.1.
Time Frame: Every 3 cycles during treatment period and at least 4 weeks after the first observation of a complete or partial response assessed up to approximately 55.9 months. The average study treatment time was 16.4 months.
Population: Eligible participants who received any amount of protocol therapy
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Ribociclib and Letrozole: Ribociclib 600 mg administered orally daily for 21 days followed by 7 days off in 28-day treatment cycle in combination with Letrozole 2.5 mg administered orally daily for 28 days.
Arm/Group | Ribociclib and Letrozole
Number analyzed (Participants) | 49
Percentage of participants | 30.6 [19.9 to 43.2]

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants in the analysis population who achieved a complete response, partial response, or stable disease, as assessed by RECIST 1.1.
Time Frame: as for outcome 1
Population: Eligible participants who received any amount of protocol therapy.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Ribociclib and Letrozole: Ribociclib 600 mg administered orally daily for 21 days followed by 7 days off in 28-day treatment cycle plus Letrozole 2.5 mg administered orally daily for 28 days.
Arm/Group | Ribociclib and Letrozole
Number analyzed (Participants) | 49
Percentage of participants | 83.7 [72.5 to 91.6]

3. Secondary Outcome: Incidence of Adverse Events (Grade 3 or Higher)
Description: Number of participants who experienced at least one adverse event of grade 3 or higher. Adverse events were graded and categorized using CTCAE v5.0.
Time Frame: During treatment period and up to 30 days after discontinuation of protocol therapy. The median duration of study treatment was 10 months with a range from 3 days to 55.9 months.
Population: Eligible participants who received any amount of protocol therapy.
Measure: Number; unit: participants
Arm/Group | Ribociclib and Letrozole
Number analyzed (Participants) | 49
participants
  Blood and lymphatic system disorders | 2
  Cardiac disorders | 1
  Eye disorders | 1
  Gastrointestinal disorders | 15
  General disorders and administration site conditions | 2
  Infections and infestations | 6
  Injury, poisoning and procedural complications | 2
  Investigations | 25
  Metabolism and nutrition disorders | 6
  Musculoskeletal and connective tissue disorders | 3
  Nervous system disorders | 2
  Psychiatric disorders | 1
  Renal and urinary disorders | 3
  Respiratory, thoracic and mediastinal disorders | 3
  Skin and subcutaneous tissue disorders | 1
  Vascular disorders | 5

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from study entry to the first documented disease progression, or death from any cause, whichever occurs first. Disease progression was assessed by RECIST 1.1.
Time Frame: From date of protocol entry to date of first documented progression or death assessed up to approximately 55 months
Population: Eligible participants who received any amount of protocol therapy
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ribociclib and Letrozole
Number analyzed (Participants) | 49
Months | 14.5 [10.1 to 28.8]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from study entry to death from any cause.
Time Frame: From date of protocol entry to date of death assessed up to approximately 62 months.
Population: Eligible participants who received any amount of protocol therapy.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ribociclib and Letrozole
Number analyzed (Participants) | 49
Months | 44.5 [31.8 to NA] — The number of events was not sufficient for the estimation of this parameter (i.e. upper limit of the CI)

6. Other Pre Specified Outcome: ER Expression
Description: Determine the expression of estrogen receptor (ER) and correlation with response and clinical benefit.
Time Frame: At time of primary and secondary outcome analysis up to 5 years.
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Mutation Analysis of Genomic Signatures
Description: Determine genomic signatures associated with response and clinical benefit of the combination of letrozole + Ribociclib
Time Frame: At time of primary and secondary outcome analysis up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: PR Expression
Description: Determine the expression of progesterone receptor (PR) and correlation with response and clinical benefit.
Time Frame: At time of primary and secondary outcome analysis up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Ki-67 Expression
Description: Determine the expression of proliferative index (ki-67) and correlation with response and clinical benefit.
Time Frame: At time of primary and secondary outcome analysis up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The time frame for adverse events was during treatment period and up to 30 days after discontinuation of protocol therapy. The median duration of study treatment was 10 months with a range from 3 days to 55.9 months. The time frame for all-cause mortality was from date of protocol entry to date of death, assessed up to approximately 62 months.
Description: Eligible participants who received any amount of protocol therapy.
Arm/Group | Ribociclib and Letrozole
All-Cause Mortality (participants affected / at risk) | 22/49
Serious Adverse Events (participants affected / at risk) | 29/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib and Letrozole (N=49)
Anemia (Blood and lymphatic system disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Eye Disorders - Other (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 6
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 5
Ileus (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Urinary Tract Infection (Infections and infestations) | 3
Small Intestine Infection (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Infections And Infestations - Other (Infections and infestations) | 1
Kidney Infection (Infections and infestations) | 1
Injury, Poisoning And Procedural Complications - O (Injury, poisoning and procedural complications) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Alcohol Intolerance (Metabolism and nutrition disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Nervous System Disorders - Other (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Suicide Attempt (Psychiatric disorders) | 1
Renal Calculi (Renal and urinary disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib and Letrozole (N=49)
Anemia (Blood and lymphatic system disorders) | 25
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 4
Palpitations (Cardiac disorders) | 3
Sinus Bradycardia (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 4
Cardiac Disorders - Other (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 1
Chest Pain - Cardiac (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Eye Disorders - Other (Eye disorders) | 1
Floaters (Eye disorders) | 1
Dry Eye (Eye disorders) | 2
Eyelid Function Disorder (Eye disorders) | 1
Eye Pain (Eye disorders) | 2
Blurred Vision (Eye disorders) | 9
Papilledema (Eye disorders) | 1
Watering Eyes (Eye disorders) | 5
Photophobia (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 22
Dry Mouth (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 17
Colitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 18
Stomach Pain (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Rectal Pain (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 11
Rectal Hemorrhage (Gastrointestinal disorders) | 2
Anal Fissure (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 4
Periodontal Disease (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 28
Mucositis Oral (Gastrointestinal disorders) | 11
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 2
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 7
Ascites (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 21
Gastritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Belching (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Pain (General disorders) | 7
Malaise (General disorders) | 2
Injection Site Reaction (General disorders) | 1
Flu Like Symptoms (General disorders) | 3
Fever (General disorders) | 5
General Disorders And Administration Site Conditio (General disorders) | 2
Fatigue (General disorders) | 30
Gait Disturbance (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 4
Edema Limbs (General disorders) | 6
Chills (General disorders) | 4
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 1
Allergic Reaction (Immune system disorders) | 1
Urinary Tract Infection (Infections and infestations) | 10
Thrush (Infections and infestations) | 1
Vaginal Infection (Infections and infestations) | 1
Small Intestine Infection (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Shingles (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Infections And Infestations - Other (Infections and infestations) | 8
Folliculitis (Infections and infestations) | 1
Eye Infection (Infections and infestations) | 2
Herpes Simplex Reactivation (Infections and infestations) | 1
Kidney Infection (Infections and infestations) | 1
Upper Respiratory Infection (Infections and infestations) | 3
Bacteremia (Infections and infestations) | 1
Prolapse Of Intestinal Stoma (Injury, poisoning and procedural complications) | 1
Intestinal Stoma Site Bleeding (Injury, poisoning and procedural complications) | 1
Injury, Poisoning And Procedural Complications - O (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Weight Loss (Investigations) | 7
Weight Gain (Investigations) | 3
Platelet Count Decreased (Investigations) | 8
Neutrophil Count Decreased (Investigations) | 34
Lymphocyte Count Increased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 11
Investigations - Other (Investigations) | 2
Inr Increased (Investigations) | 8
Creatinine Increased (Investigations) | 22
Cpk Increased (Investigations) | 4
Cholesterol High (Investigations) | 6
Lipase Increased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 27
Aspartate Aminotransferase Increased (Investigations) | 10
Alkaline Phosphatase Increased (Investigations) | 12
Alanine Aminotransferase Increased (Investigations) | 11
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hyperuricemia (Metabolism and nutrition disorders) | 10
Hypertriglyceridemia (Metabolism and nutrition disorders) | 9
Hyperphosphatemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hypercalcemia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 16
Alcohol Intolerance (Metabolism and nutrition disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 12
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 5
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 4
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 2
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tremor (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Stroke (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 4
Neuralgia (Nervous system disorders) | 1
Nervous System Disorders - Other (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 17
Paresthesia (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Extrapyramidal Disorder (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 10
Suicide Attempt (Psychiatric disorders) | 1
Psychiatric Disorders - Other (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 6
Urinary Tract Pain (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 8
Renal Calculi (Renal and urinary disorders) | 1
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 12
Urinary Incontinence (Renal and urinary disorders) | 2
Urinary Urgency (Renal and urinary disorders) | 4
Hematuria (Renal and urinary disorders) | 7
Glucosuria (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 7
Cystitis Noninfective (Renal and urinary disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 2
Bladder Spasm (Renal and urinary disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2
Vaginal Dryness (Reproductive system and breast disorders) | 4
Vaginal Discharge (Reproductive system and breast disorders) | 1
Uterine Pain (Reproductive system and breast disorders) | 1
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 3
Pelvic Pain (Reproductive system and breast disorders) | 5
Vaginal Pain (Reproductive system and breast disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 7
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 5
Nail Changes (Skin and subcutaneous tissue disorders) | 2
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 12
Thromboembolic Event (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 11
Hot Flashes (Vascular disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03673124/Prot_SAP_000.pdf